CLINICAL TRIAL: NCT05412459
Title: SPECT Imaging of Human Epidermal Growth Factor Receptor 2 (HER2) Using 99mTc-DARPinG3 in HER2-positive Breast Cancer Patients in Dynamic of Chemo+Targeted Therapy
Brief Title: 99mTc-DARPinG3-based HER2 Expression Molecular Imaging in HER2-positive Breast Cancer During Chemo+Targeted Therapy
Status: Completed | Type: Observational
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Collaborators: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: 99mTc-DARPinG3
Record Dates: First submitted 2022-06-02; First posted 2022-06-09 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2022-06

CONDITIONS: HER2-positive Breast Cancer; Female
Keywords: 99mTc-DARPinG3; Breast Cancer; HER2 expression; chemotherapy and targeted therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor biopsies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The tested injected doses of 99mTc-DARPinG3 3000 μg (SPECT): Maximum (15) evaluable subjects with HER2-positive status in primary tumour before, after 2 and 4 courses of chemo+targeted therapy have to be enrolled in the study.
  Subjects withdrawn from the study for any reason will be replaced.
  Interventions: Drug: 99mTc-DARPinG3

INTERVENTIONS:
Drug: 99mTc-DARPinG3 — Diagnostic test (99mTc-DARPinG3-based SPECT) is used for the assessment of the effect of anticancer therapy.
  Other Names: Diagnostic injection of 99mTc-DARPinG3.

SUMMARY:
An open-label, single center study with 99mTc-DARPinG3 SPECT and biopsies of primary tumour in HER2-positive Breast Cancer in dynamic of chemo+targeted therapy, where the primary endpoint of the study is to find out the correlation between the HER2 expression measured by 99mTc-DARPin G3 SPECT and standard histopathology from primary tumor in dynamic of chemo+targeted therapy.

DETAILED DESCRIPTION:
none Methodology: Open-label, exploratory, single center study. The subjects will receive a single injection of the labelled tracer.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is > 18 years of age;
2. Diagnosis of primary breast cancer with tumour size ≥ 20 mm and with possible lymph node metastases;
3. Availability of results from HER2 status previously determined on material from the primary tumor: HER2-positive, defined as a DAKO HercepTest™ score of 3+ or FISH positive;
4. In neoadjuvant all patients should receive standard chemo-targeted therapy according to the DCH+P (docetaxel + carboplatin+ trastuzumab+ pertuzumab) scheme;
5. Injection of 99mTc-DARPinG3 at the dosage 3000 µg before and after 2 and 4 courses of chemo+targeted therapy in each HER2-positive breast cancer patient;
6. Biopsies should be performed in all patients HER2-positive breast cancer patients before and after 2 and 4 courses of chemo+targeted therapy with evaluation of HER2 expression;
7. Hematological, liver and renal function test results within the following limits:

   * White blood cell count: > 2.0 x 109/L
   * Hemoglobin: > 80 g/L
   * Platelets: > 50.0 x 109/L
   * ALT, ALP, AST: =< 5.0 times Upper Limit of Normal
   * Bilirubin =< 2.0 times Upper Limit of Normal
   * Serum creatinine: Within Normal Limits
8. A negative pregnancy test for all patients of childbearing potential. Sexually active women of childbearing potential participating in the study must use a medically acceptable form of contraception for at least 30 days after study termination;
9. Subject is capable to undergo the diagnostic investigations to be performed in the study;
10. Informed consent

Exclusion Criteria:

1. Second, non-breast malignancy
2. Active current autoimmune disease or history of autoimmune disease
3. Active infection or history of severe infection within the previous 3 months (if clinically relevant at screening) 4. Known HIV positive or chronically active hepatitis B or C
4. Administration of other investigational medicinal product within 30 days of screening
5. Ongoing toxicity > grade 2 from previous standard or investigational therapies, according to US National Cancer Institute's

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females
Study Population: Breast cancer female patients.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
SPECT/CT-based 99mTc-DARPinG3 uptake value in primary tumor (standardized uptake value (SUV)) | 4 hours
  SPECT/CT-based 99mTc-DARPinG3 uptake value in primary tumor lesions (SUV) of 99mTc-DARPinG3 focal uptake coinciding with tumor lesions will be assessed using SPECT/CT at 4 hours after injection and measured in counts and SUV before and after 2 and 4 courses of chemo+targeted therapy
SPECT-based tumor-to-background ratio (conventional units) | 4 hours
  The SPECT-based tumor-to-background ratio will be calculated as follows: the value of 99mTc-DARPinG3 uptake coinciding with primary tumor lesions (SUV) will be divided by the value of 99mTc-DARPinG3 uptake coinciding with the regions without pathological findings (SUV) before and after 2 and 4 courses of chemo+targeted therapy

SECONDARY OUTCOMES:
Tumor-to-background ratio 99mTc-DARPinG3 SPECT versus immunohistochemical study | 4 hours
  Comparison of the 99mTc-DARPinG3 accumulation (SUV or count-to-background ratio) in primary tumour with the results of morphological and immunohistochemical studies (score from 1 to 3) before and after 2 and 4 courses of chemo+targeted therapy

CONTACTS AND LOCATIONS:
Overall Officials: Olga Bragina, MD, Dsc, Principal Investigator — Tomsk NRMC
Locations (2):
- Russia (2):
  - Tomsk NRMC, Tomsk
  - TomskNRMC, Tomsk